CLINICAL TRIAL: NCT05017415
Title: What is the Difference in the Applicability of the Uroflowmetry Between Children with Cerebral Palsy (CP) with Lower Urinary Tract Symptoms (LUTS) and Without Lower Urinary Tract Symptoms (LUTS)
Brief Title: Applicability of Uroflowmetry in Children with Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: BC-9774
Record Dates: First submitted 2021-08-16; First posted 2021-08-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Palsy; Lower Urinary Tract Symptoms
Keywords: cerebral palsy; lower urinary tract symptoms; incontinence; uroflow measurement
MeSH Terms: conditions — Cerebral Palsy; Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: Children will be randomised in two groups, with evaluation with a standard toilet seat or a toilet seat with decreased hip angle.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard toilet chair (hip angle 90°) (Experimental): uroflow measurement with subsequent post void residual measurement, conducted on a standard toilet chair.
  Interventions: Device: uroflow measurement; Device: Bladder ultrasound
- Toilet chair with decreased hip angle (Experimental): uroflow measurement with subsequent post void residual measurement, conducted on a toilet chair with decreased hip angle.
  Interventions: Device: uroflow measurement; Device: Bladder ultrasound

INTERVENTIONS:
Device: uroflow measurement — Non-invasive urodynamic measurement wireless uroflowmeter UROCAP™ IV, Goby System Laborie
  Other Names: uroflowmetry
Device: Bladder ultrasound — Ultrasound of post void residual urine bladderscan CUBEscan BioCon 700
  Other Names: US

SUMMARY:
Until now, the use of invasive urodynamics with use of catheters is still the gold standard for lower urinary tract evaluation in subjects with CP. This suggests a psychological and physical impact of invasive urodynamics in subjects with CP and further demonstrates the need to avoid standard use of invasive urodynamics in children and adults with CP.

The current study will evaluate usefulness of uroflowmetry, correlation between uroflowmetry parameters and different lower urinary tract symptoms will be investigated. Secondly, results of uroflowmetry indicating possible vulnerability of the upper urinary tract will be defined.

DETAILED DESCRIPTION:
A cross-sectional case-control study comparing children with CP and LUTS and children with CP without LUTS will be conducted with the primary objective to investigate correlation between uroflowmetry parameters and different LUTS.

Children will be evaluated with uroflowmetry and subsequent post void residual measurement and the validated vancouver symptom score for dysfunctional elimination syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cerebral palsy
* Dutch or French speaking child and parent

Exclusion Criteria:

* History of urological surgery

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Amount of pathological uroflow patterns - Qualitative assessment | During cross-sectional testing
  Interpretation by pediatric urologist following ICCS classification Measured during uroflowmetry
Amount of pathological uroflow patterns - Quantitative assessment | During cross-sectional testing
  Interpretation using Flow index methodology Measured during uroflowmetry
Maximal flow | During cross-sectional testing
  Measured during uroflowmetry Qmax (mililitres/seconds

SECONDARY OUTCOMES:
Influencing factors for uroflow measurement | During cross-sectional testing
  * Functional impairment of the child
  * hip angle
  * Vancouver symptom score for dysfunctional elimination syndrome
Voided volume | During cross-sectional testing
  Measured during uroflowmetry mililitres Percentage of expected bladder capacity
Post void residual urine | During cross-sectional testing
  Measured with CUBEscan BioCon 700 mililiters Percentage of voided volume

CONTACTS AND LOCATIONS:
Overall Officials: Bieke Samijn, dr., Principal Investigator — Ghent University Hospital/Ghent University
Locations (1):
- Ghent University Hospital, Ghent, Flanders, Belgium